CLINICAL TRIAL: NCT04606485
Title: The Effect On Gastrointestinal System Functions, Pain And Anxiety Of Acupressure Applied Following Laparoscopic Cholecystectomy Operation: A Randomised, Placebo-Controlled Study
Brief Title: Does Acupressure Affect Gastrointestinal Function, Pain and Anxiety?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Di̇lek Soylu, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Interventional
Record Dates: First submitted 2020-10-13; First posted 2020-10-28 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Gastrointestinal Dysfunction; Anxiety; Pain, Postoperative
Keywords: Acupressure; Gastrointestinal Dysfunction; Anxiety; Pain
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative; Pain | interventions — Acupressure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Acupressure was applied to both the intervention and placebo groups, by a single nurse researcher, trained in the application of acupressure. The nurse had received a certificate for attendance of an acupressure course which included theoretical and practical lessons for specialization on the subject of acupressure. Patients in the placebo group were unaware of their group. Patients were isolated from others by using acupressure in single rooms or by using a curtain around the bed. Thus, it was ensured that the patients were not affected by each other.
  Another nurse researcher blinded to the groups collected the data. The statistics specialist who analysed and reported the data was also blinded to the groups. Analysis and reporting were also defined as groups 1 and 2. Thus the 3-way blinded technique was used in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Since acupressure administration was reported to have placebo effects, a placebo group was used to investigate the true effect of acupressure use. The application of placebo may consist of moderate pressure on an incorrect acupuncture point or a light touch on a real acupuncture point. This will allow us to determine the contribution of the placebo effect resulting from direct human contact and interaction in the light touch group.
  At postoperative 0, 4, and 8 hours, a light touch was applied to the ST25 (Stomach Meridian 25th point), CV12 (Conception Vessel Meridian 12th point), TH6 (Triple Heater Meridian 6th point) and HT7 (Shenmen point points) for one second. No patients experienced pain or a feeling of pressure.
  Interventions: Other: Acupressure
- Experimental group (Experimental): As invasive acupuncture may cause hematoma and the wristband method of non-invasive acupressure may cause patient discomfort, itching, swelling of the wrist, and skin destruction, manual acupressure was applied in this study to reduce the risk of complications to a minimum.
  The frequency and duration of the application of acupressure was decided from a scan of literature and expert opinion. The first acupressure session was applied in the first postoperative hour immediately after routine treatment and care of the patients who came to the ward from the recovery unit. Acupressure by applying pressure with the thumbs for a total of 12 mins, as 3 mins at each of the ST25, CV12, TH6 and HT7 acupuncture points, was performed at 0, 4 and 8 hours postoperatively. The acupuncture points were determined using the measurements of the patient's own fingers.
  Interventions: Other: Acupressure

INTERVENTIONS:
Other: Acupressure — Acupressure is accepted as a non-invasive application that can easily be applied by trained nurses, which increases the quality of the medical care administered and contributes to physical and psychological recovery.

SUMMARY:
The aim of this randomised, placebo-controlled, 3-way blinded study was to determine the effect on GIS symptoms, pain and anxiety of acupressure applied for a total of 12 mins, as 3 mins at each of the ST25, CV12, TH6 and HT7 acupuncture points, at 0, 4 and 8 hours after laparoscopic cholecystectomy operation. The research data were collected using a patient data collection form, the Numeric Pain Intensity Scale and the State-Trait Anxiety Inventory. The patients were evaluated in respect of the time to first flatus and defecation, pain and the State-Trait Anxiety points at 0, 4, and 8 hours postoperatively.

DETAILED DESCRIPTION:
Together with technological advances in the field of healthcare, there is currently a greater preference for the laparoscopic cholecystectomy procedure, as length of hospital stay is shorter, workforce loss is lower, good cosmetic results are obtained and postoperative patient satisfaction is higher, when compared to open cholecystectomy.

One of the basic factors affecting the patient is the anesthesia applied in the laparoscopic surgical approach. Following general anaesthesia, metabolic activity slows and gastrointestinal system (GIS) movements are reduced. In addition, by increasing intra-abdominal pressure, the gas insufflation applied to the peritoneal cavity in laparoscopic surgery, reduces blood flow in the stomach and small and large intestines. As a result of this reduced blood flow, ischemia and dysfunction in the intestines may cause ileus symptoms to emerge. Pain occuring as a response to surgical stress causes a decrease in intestinal motility. If pain is not brought under control postoperatively, nausea, vomiting, constipation and ileus may occur.

Preoperative anxiety has been reported to be associated with postoperative pain, cognitive disorders and delayed healing. Stress reaction, surgical intervention to the abdominal region, trauma, postoperative pain, and the use of anaesthetic and narcotic agents are among the factors causing the development of GIS problems. An increase in sympathetic activity which occurs in the stress reaction and the use of general/narcotic anaesthesia reduce gastrointestinal motility. Pharmacological treatments are applied to improve GIS functions. It has been reported that intravenous infusion of lidocaine in the perioperative period provides a faster recovery of bowel functions. Postoperative gastrointestinal dysfunction is usually treated using alvimopan, but the drug used has side effects such as nausea and vomiting. Postoperative pain and nausea-vomiting are common complaints after laparoscopic cholecystectomy, despite the use of multimodal analgesia consisting of dexamethasone, opioids, nonsteroidal anti-inflammatory drugs and local anesthetics used in the perioperative period. In addition, of the nursing applications used, the application of acupressure is of benefit. Acupressure is accepted as a non-invasive application that can easily be applied by trained nurses, which increases the quality of the medical care administered and contributes to physical and psychological recovery. In studies of acupressure applied for the recovery of GIS functions, it has been reported that acupressure can be applied as non-invasive nursing care which improves postoperative ileus symptoms.

In a study by Chao et al, acupressure applied after abdominal surgery was reported to improve gas output, shorten the time to oral nutritional intake, and improve ileus symptoms. Acupressure applied to the P6 point following appendectomy decreased the frequency of vomiting. In another study, acupressure was determined to be effective in improving GIS movement. Acupressure improved intestinal functions but stated that more experimental studies were needed.

It is recommended to teach the use of acupuncture warning devices to patients with post-operative nausea, vomiting and anxiety problems. However, there is no definitive evidence as to when, how and for how long acupressure should be administered. Moreover, studies conducted by nurses on this subject are limited and studies with high evidence value are needed. As a result of our literature review, the effect of acupressure applied to ST25, CV12, TH6 and HT7 on bowel movements, first flatus and defecation time, pain and anxiety after laparoscopic cholecystectomy was not investigated. Therefore, our study was carried out to evaluate the effect of acupressure applied to patients after laparoscopic cholecystectomy on GIS functions, pain and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Able to understand the information given
* Willing to receive acupressure
* No lesions or wounds in the areas where acupressure was to be applied
* Operated on under general anaesthesia pulse, blood pressure, body temperature and oxygen saturation values within normal range during the operation
* No failure or disorder developing intraoperatively or postoperatively related to fluid-electrolyte balance, acid-base balance, or tissue perfusion.

Exclusion Criteria:

* American Society of Anaesthesiologists (ASA) physical status IV
* A requirement for simultaneous combined surgery,
* A need for postoperative fasting according to the preoperative evaluation or intraoperative findings (eg, panperitonitis with intraperitoneal abscess)
* Patients with a cardiac pacemaker
* A history of syncope or seizures
* Pregnant or lactating women
* The presence of any disease related to bleeding or a clotting disorder
* Patients who were unwilling to participate in the research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Change in the first flatus process according to the information received from the patient | Postoperative 0 and 72 hours
  First flatus hour is validated, the patient was questioned about the time of flatus output. The hour reported by the patient was evaluated as the time of first flatus. Change=(Postoperative 0 and 72 hours).
Change in the first gaits output process according to the information received from the patient | Postoperative 0 and 72 hours
  First gaits output is validated, the patient was questioned about the time of gaits output. The hour reported by the patient was evaluated as the time of first gaits.Change=(Postoperative 0 and 72 hours).
Change from Baseline in Pain on The Numeric Pain Intensity Scale (NAS) at postoperative 0, 4 and 8 hours. | Pre-acupressure, postoperative 0, 4 and 8 hours
  NAS is a single dimension, subjective scale, consisting of a horizontal line, marked at equal intervals from 0-10, where 0= no pain and 10= intolerable pain. The scores were evaluated as 1-3 represents mild pain, 4-6 moderate pain, and 7-10 severe pain. The patients were instructed to mark the number best reflecting the level of pain felt.It was evaluated 4 times in total before acupressure, at the postoperative 0, 4 and 8 hours after the acupressure application. Change=(pre-acupressure score- postoperative 0, 4 and 8 hours scores).
Change from Baseline The State-Trait Anxiety Inventory (SAI) at pre-acupressure and postoperative 8 hour | Pre-acupressure and postoperative 8 hour
  The State-Trait Anxiety Inventory was developed by Spielberger in 1964 and was adapted to Turkish by Öner and LeCompte. The scale, which is self-reported and consists of short statements, measures the levels of anxiety of both patients and healthy individuals. The State Anxiety Inventory (SAI) provides information about how the individual feels at that time, and the Trait Anxiety Inventory (TAI) about how they have felt in the last 7 days.
  The constant value is 50 for the SAI and 35 for the TAI. The most recently obtained value constitutes the anxiety points, in a maximum range of 20-80, with high scores indicating a high level of anxiety. Change= (Pre-acupressure score and postoperative 8 hour score).

SECONDARY OUTCOMES:
Change from Baseline in Nause on The Nause Intensity Scale (VAS) at pre-acupressure, postoperative 0, 4 and 8 hours. | Pre-acupressure, postoperative 0, 4 and 8 hours
  A 10 cm scale, marked in cm, where 0= no nausea and 10= very severe nausea was used and each patient was instructed to mark the greatest severity of nausea that they had felt on the scale. It was evaluated 4 times in total before acupressure, at the postoperative 0, 4 and 8 hours after the acupressure application. Change=(pre-acupressure score- postoperative 0, 4 and 8 hours score).
Change from Baseline in intestinal sounds at pre-acupressure, postoperative 0, 4 and 8 hours. | Pre-acupressure, postoperative 0, 4 and 8 hours
  Intestinal sounds were listened to with the same stethoscope, by dividing the abdomen into 4 quadrants and evaluating each quadrant. A time of one minute was set on a chronometer for each evaluation, and the number of the intestinal sounds in one minute were counted and recorded. It was evaluated 4 times in total before acupressure, at the postoperative 0, 4 and 8 hours after the acupressure application. Change=(pre-acupressure number- postoperative 0, 4 and 8 hours numbers).

CONTACTS AND LOCATIONS:
Overall Officials: Di̇lek Soylu, Principal Investigator — Kahramanmaras Sutcu Imam universty
Locations (1):
- Di̇lek Soylu, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Our study has not been published yet

REFERENCES:
- [Result] Abadi F, Shahabinejad M, Abadi F, Kazemi M. Effect of Acupressure on Symptoms of Postoperative Ileus After Cesarean Section. J Acupunct Meridian Stud. 2017 Apr;10(2):114-119. doi: 10.1016/j.jams.2016.11.008. Epub 2016 Dec 27. PMID 28483182
- [Result] Chao HL, Miao SJ, Liu PF, Lee HH, Chen YM, Yao CT, Chou HL. The beneficial effect of ST-36 (Zusanli) acupressure on postoperative gastrointestinal function in patients with colorectal cancer. Oncol Nurs Forum. 2013 Mar;40(2):E61-8. doi: 10.1188/13.ONF.E61-E68. PMID 23448746
- [Result] Adib-Hajbaghery M, Etri M, Hosseainian M, Mousavi MS. Pressure to the p6 acupoint and post-appendectomy pain, nausea, and vomiting: a randomized clinical trial. J Caring Sci. 2013 Jun 1;2(2):115-22. doi: 10.5681/jcs.2013.014. eCollection 2013 Jun. PMID 25276717
- [Result] Chen LL, Hsu SF, Wang MH, Chen CL, Lin YD, Lai JS. Use of acupressure to improve gastrointestinal motility in women after trans-abdominal hysterectomy. Am J Chin Med. 2003;31(5):781-90. doi: 10.1142/S0192415X03001466. PMID 14696681

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT04606485/Prot_SAP_ICF_000.pdf